CLINICAL TRIAL: NCT01127412
Title: Early Obesity Intervention Program Within GECKO Drenthe; a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: P.J.J. Sauer MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EOIP-GECKO
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Overweight; Physical Activity
Keywords: overweight; physical activity; infancy; body composition; motor development; motor activity
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity stimulating program (Active Comparator): Advices to stimulate motor activity and motor development at the age of two weeks, two months, four months, eight months and eleven months
  Interventions: Behavioral: Physical activity stimulating program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity stimulating program
  Arms: Physical activity stimulating program

SUMMARY:
The purpose of this study is to investigate whether stimulating physical activity during the first year of life influences growth and body composition, and stimulates motor activity and motor development

ELIGIBILITY:
Inclusion Criteria:

* date of birth (December 2006-February 2008)
* area of living (around Meppel and Hoogeveen in the province of Drenthe, one of the Northern provinces of the Netherlands)

Exclusion Criteria:

* Children under care of child physiotherapists will be excluded from the program

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Growth | Regularly during the first year of life, at 2.5 years of age
  Weight, length
Body composition | Regularly during the first year of life, at 2.5 years of age
  Waist circumference, Hip circumference, Skin fold thickness, Bioelectrical impedance analyses (BIA)

SECONDARY OUTCOMES:
Motor activity | At the age of 5 months, 8 months and 2.5 years of age
  Accelerometer
Motor development | At the age of 5 months, 8 months and 2.5 years of age
  Albertha Infant Motor Scale, Bayley Scales of Infant and Toddler Development